CLINICAL TRIAL: NCT03347708
Title: A Prospective, Randomized, Double-Blinded, Vehicle- and Placebo-Controlled, Multicenter Study to Evaluate the Safety and Preliminary Efficacy of IDCT in Subjects With Single-Level, Symptomatic Lumbar Intervertebral Disc Degeneration
Brief Title: Study to Evaluate the Safety and Preliminary Efficacy of IDCT, a Treatment for Symptomatic Lumbar Intervertebral Disc Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DiscGenics, Inc. (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DGX-A01
Record Dates: First submitted 2017-11-01; First posted 2017-11-20 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-11

CONDITIONS: Degenerative Disc Disease
Keywords: Lumbar disc degeneration; Low back pain; Intervertebral disc degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain | interventions — Saline Solution; Sodium Chloride; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- High Dose IDCT (Experimental): Single intradiscal injection with High Dose IDCT (9M cells).
  Interventions: Biological: IDCT
- Low Dose IDCT (Experimental): Single intradiscal injection with Low Dose IDCT (3M cells).
  Interventions: Biological: IDCT
- Saline (Placebo Comparator): Single intradiscal injection with saline solution.
  Interventions: Drug: Saline Solution
- Sodium Hyaluronate Vehicle (Placebo Comparator): Single intradiscal injection with Sodium Hyaluronate Vehicle.
  Interventions: Drug: Sodium Hyaluronate

INTERVENTIONS:
Biological: IDCT — Discogenic Cells + Sodium Hyaluronate Vehicle
  Other Names: Progenitor Cells, Stem Cells, Allogeneic Cell Therapy
  Arms: High Dose IDCT; Low Dose IDCT
Drug: Saline Solution — Sodium Chloride Solution
  Other Names: Saline injection, Placebo control
  Arms: Saline
Drug: Sodium Hyaluronate — Sodium Hyaluronate Vehicle
  Other Names: Sodium Hyaluronate injection, Hyaluronate Acid, Sodium Hyaluronate Solution Vehicle control
  Arms: Sodium Hyaluronate Vehicle

SUMMARY:
The purpose of this study is to compare the safety and preliminary efficacy of intradiscal injections of two doses of IDCT (Discogenic Cells + Sodium Hyaluronate vehicle) and two controls (saline, Sodium Hyaluronate vehicle) in subjects with chronic low back pain due to Degenerative Disc Disease (DDD) at one lumbar level from L3 to S1.

DETAILED DESCRIPTION:
This is a Phase I, first-in-human, randomized, double-blind, vehicle and placebo-controlled, parallel-group, multi-center study in subjects with single-level, symptomatic lumbar intervertebral disc degeneration (>6 months) and unresponsive to conservative therapy for at least 3 months. The study will compare single intradiscal injections of high and low dose IDCT with two control groups (saline, Sodium Hyaluronate).

8 study visits will be completed by all subjects; screening, day 1 (injection day), week 4, week 12, week 26, week 52, week 72 and week 104. The subject will be assessed for safety and efficacy utilizing VAS and ODI questionnaires alongside radiographic evaluations. The study will have a 1 year follow-up and a 1 year extension period (total 2 years).

ELIGIBILITY:
Inclusion Criteria: The subject must have:

1. Diagnosis of early to moderate degenerative disc disease (DDD), Modified Pfirrmann Grade 3-7.
2. Chronic low-back pain for at least 6 months prior to screening; unresponsive to at least 3 months of conservative care.
3. Low-back pain of 40 to 90 mm on the VAS and ODI score of 30 to 90.

Exclusion Criteria: The subject is excluded if he/she has:

1. Symptomatic involvement of more than one lumbar disc.
2. Other persistent pain/nerve issues including, for example, radiculopathy, leg pain, cauda equine syndrome, etc.
3. Fracture of the spine, previous lumbar spine surgery or previous treatment of the target disc.
4. Evidence of dynamic instability on lumbar flexion-extension radiographs.
5. Grade 2 or higher spondylolisthesis at the target disc, lumbar spondylitis or other undifferentiated spondyloarthropathy, or Type III Modic changes around the target disc.
6. Clinical suspicion of a full thickness annular tear at the target disc or other abnormal disc morphology.
7. Clinical suspicion of facet pain as primary pain generator.
8. Subjects who test positive for communicable disease, have significant systemic disease, or are prone to infection.
9. Patients who are deemed unsuitable for clinical study participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Safety as measured by number of Adverse Events | 2 Years
  To evaluate the safety and tolerability of a single injection of IDCT in subjects with single-level, symptomatic early to moderate lumbar intervertebral disc degeneration as measured by the incidence of grade 2 or greater AEs and SAEs observed from Day 1 to week 104
Efficacy (Pain) | 1 Year
  Evaluate the effect of IDCT on pain as measured by a 0-100mm Visual Analogue Scale (VAS). 0: no pain, 100: worst pain imaginable.

SECONDARY OUTCOMES:
Disability | 2 Years
  Evaluate the effect of IDCT on disability as measured by the Oswestry Disability Index (ODI). Score of 0%: no disability, score of 100%: severely disabled

OTHER OUTCOMES:
Exploratory | 2 Years
  Imaging parameters will be evaluated via radiological evaluations

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - UC San Diego CIRM Alpha Stem Cell Clinic, San Diego, California
  - Source Healthcare, Santa Monica, California
  - Otrimed, Edgewood, Kentucky
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Orthopedic Center of St. Louis, Chesterfield, Missouri
  - Ainsworth Institute of Pain Management, New York, New York
  - Carolina Neurosurgery & Spine Associates, Charlotte, North Carolina
  - Clinical Investigations, LLC, Edmond, Oklahoma
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Semmes Murphey, Memphis, Tennessee
  - Physicians' Research Options, LLC, Draper, Utah
  - Virginia iSpine, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gornet MF, Beall DP, Davis TT, Coric D, LaBagnara M, Krull A, DePalma MJ, Hsieh PC, Mallempati S, Schranck FW, Kelly C, Foley KT. Allogeneic Disc Progenitor Cells Safely Increase Disc Volume and Improve Pain, Disability, and Quality of Life in Patients With Lumbar Disc Degeneration-Results of an FDA-Approved Biologic Therapy Randomized Clinical Trial. Int J Spine Surg. 2024 Jul 4;18(3):237-248. doi: 10.14444/8609. PMID 38925869
- [Derived] Silverman LI, Dulatova G, Tandeski T, Erickson IE, Lundell B, Toplon D, Wolff T, Howard A, Chintalacharuvu S, Foley KT. In vitro and in vivo evaluation of discogenic cells, an investigational cell therapy for disc degeneration. Spine J. 2020 Jan;20(1):138-149. doi: 10.1016/j.spinee.2019.08.006. Epub 2019 Aug 20. PMID 31442616
- See also: Related Info — http://www.discgenics.com